CLINICAL TRIAL: NCT02913443
Title: A Multi-Center, Open Label, Phase I, Dose Finding and Expansion Study of RO7051790 Administered Orally in Patients With Relapsed, Extensive-Stage Disease Small Cell Lung Cancer (ED SCLC)
Brief Title: A Dose Finding and Expansion Study of RO7051790 Administered Orally in Participants With Relapsed, Extensive-Stage Disease Small Cell Lung Cancer (ED SCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NP39148; 2016-001942-25 (EudraCT Number)
Record Dates: First submitted 2016-09-16; First posted 2016-09-23 (Estimated); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

ARMS (4):
- Introductory Cohort - 400 μg RO7051790 (Experimental): Introductory cohort to ensure participant safety, prior to the dose escalation study. 400 μg of RO7051790 was administered to two (2) participants followed by a 21-day DLT observation period.
  Interventions: Drug: RO7051790
- Dose Escalation - 1000 μg RO7051790 (Experimental): 1000 μg of RO7051790 was administered to six (6) participants once every 3 weeks (Q3W).
  Interventions: Drug: RO7051790
- Dose Escalation - 1300 μg RO7051790 (Experimental): 1300 μg of RO7051790 was administered to seven (7) participants once every 3 weeks (Q3W).
  Interventions: Drug: RO7051790
- Dose Escalation - 1900 μg RO7051790 (Experimental): 1900 μg of RO7051790 was administered to three (3) participants once every 3 weeks (Q3W).
  Interventions: Drug: RO7051790

INTERVENTIONS:
Drug: RO7051790 — RO7051790 will be given orally. Treatment will be continued until disease progression/treatment failure, unacceptable toxicity, or study discontinuation.

SUMMARY:
This is a Phase I, open-label, multicenter study designed to assess the safety and tolerability of RO7051790 in participants with relapsed ED SCLC. This dose escalation and expansion study plans to determine the maximum tolerated dose and/or optimal biological dose as a recommended Phase 2 dose for RO7051790, based on the safety, tolerability, pharmacokinetic and pharmacodynamic profiles observed after oral administration of RO7051790.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy greater than or equal to (>=) 12 weeks
* Participants must have histologically or cytologically confirmed diagnosis of SCLC
* Participants must have recurrent or refractory disease after receiving at least one prior platinum-containing chemotherapy regimen, or standard therapy is refused or not suitable. For participants in Canada: participants should also not be suitable for treatment with topotecan hydrochloride
* Acute toxicities from any prior treatment, surgery, or radiotherapy must be National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03 Grade less than or equal to (<=) 1
* Measureable disease per RECIST v1.1 prior to administration of study medication
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Adequate bone marrow function
* Adequate renal function
* Participant must be able to swallow and retain orally administered study treatment
* Women of childbearing potential and men should agree to use an effective form of contraception and to continue its use for the duration of study treatment and for a period of time after the last dose of study treatment

Exclusion Criteria:

* Active malignancy other than SCLC within the previous 5 years
* Participants who have received radiotherapy less than 2 weeks prior to first dose of study medication
* Surgical procedure or clinically significant trauma within 2 weeks of first dose of study treatment
* Treatment with any investigational agent <=3 weeks prior to first dose of study treatment
* Participants with gastrectomy or pre-existing gastrointestinal disorders that may interfere with the proper absorption of the drug(s), as per conclusion of the clinical Investigator
* Participants medicated with anti-depressants reported to have lysine-specific histone demethylase 1A (KDM1A)/lysine (K)-specific demethylase 1A (LSD1) inhibitory activity (such as tranylcypromine or phenelzine) within 28 days of treatment start
* History of allergic reactions attributed to components of the formulated product(s)
* History of seizure disorders
* Participants with untreated central nervous system metastases, or history of previously treated disease. Participants must have stable hematological parameters, satisfying eligibility, platelet count must be stable for >=2 weeks prior to study drug administration
* Participants who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study
* Participants with evidence of electrolyte imbalance
* Participants who are pregnant or breastfeeding
* Participants who refuse to potentially receive blood products and/or have a hypersensitivity to blood products
* Participants with known bone marrow disorders which may interfere with bone marrow recovery or participants with delayed recovery from prior chemoradiotherapy
* Participants with known coagulopathy, platelet disorder or history of non-drug-induced thrombocytopenia
* Hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV)-positive participants with active infection
* Use of strong Cytochrome P450 3A4 (CYP3A4) inducers while on study medication
* Participants with abnormal hepatic function
* Participants with history of clinically significant bleeding, specifically any history of intracranial hemorrhage/hemorrhagic cardiovascular accident (CVA), or participants with gastrointestinal bleeding within the 12 months prior to study entry
* Participants receiving therapeutic anti-coagulation or anti-platelet (anti-aggregant) therapies, except for therapeutic enoxaparin or low dose aspirin. Use of subcutaneous heparin prophylaxis, including low molecular weight heparin is also permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2017-10-24 (Actual); Study Completion 2017-10-24 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events | Baseline up to approximately 18 weeks
Number of Participants with Dose-Limited Toxicities (DLTs) | First treatment cycle (21 days)
  DLTs were to be assessed based on the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03. DLTs were at least possibly related to RO7051790 and had to meet any one of the following criteria: Grade≥4 neutropenia lasting >7 days; Grade 4 thrombocytopenia; Grade 3 thrombocytopenia with bleeding; Grade≥4 anemia; Febrile neutropenia; Grade≥3 elevation in serum hepatic transaminase lasting >7 days; Grade≥3 elevation of serum bilirubin; and Grade≥3 non-hematologic, non-hepatic adverse event (with few exceptions).

SECONDARY OUTCOMES:
Percentage of Participants with Best Confirmed Overall Response | Time from first study treatment to the time of progression or death from any cause, whichever occurs first (Assessed every 6 weeks up to approximately 18 weeks)
  Best Confirmed Overall Response was evaluated according to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1). Complete Response (CR) included the disappearance of all target lesions; Partial Response (PR) was at least a 30% decrease in the sum of diameters of target lesions; Progressive Disease (PD) was at least a 20% increase in the sum of diameters of target lesions; and Stable Disease (SD) was neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Percentage of Participants with Objective Response According to RECIST | Time from first study treatment to the time of progression or death from any cause, whichever occurs first (assessed every 6 weeks up to approximately 18 weeks)
  Objective response was defined as the percentage of participants with a Complete Response (CR) or Partial Response (PR) as defined by the Response Evaluation Criteria in Solid Tumors (RECIST). CR was defined as the disappearance of all target lesions; PR was defined as a 30% decrease in sum of longest diameter of target lesions.
Duration of Response According to RECIST v1.1 | Time from first occurrence of a documented objective response to the time of progression or death from any cause, whichever occurs first (assessed every 6 weeks up to approximately 18 weeks)
  Duration of response was defined as the interval between the date of the first documented response by RECIST to the date of first disease progression or death, whichever occurred earlier.
Progression-Free Survival (PFS) According to RECIST v1.1 | Time from first study treatment to the time of progression or death from any cause, whichever occurs first (assessed every 6 weeks up to approximately 18 weeks)
  Progression-free survival was defined as the time from the first administration of any study treatment to the first disease progression using RECIST or death from any cause, whichever occurred first.
Overall Survival (OS) | Time from first study treatment to death from any cause (up to approximately 12 months)
Maximum Observed Plasma Concentration (Cmax) of RO7051790 | Predose (0 hours [hrs]) on Day 1 of every cycle until end of treatment (up to 18 weeks, each cycle is 21 days); Cycles 1 and 2: 1,2,4,6,8 (only in Cycle 1) hrs postdose on Day 1 and on Days 2 (only in Cycle 1), 4, 5 (only in Cycle 1), 8,12,15,19
Minimum Observed Plasma Trough Concentration (Cmin) of RO7051790 | Predose (0 hrs) on Day 1 of every cycle until end of treatment (up to 18 weeks, each cycle is 21 days)
Time to Reach Maximum Observed Plasma Concentration (Tmax) of RO7051790 | Predose (0 hrs) on Day 1 of every cycle until end of treatment (up to 18 weeks, each cycle is 21 days); Cycles 1 and 2: 1, 2, 4, 6, 8 (only in Cycle 1) hrs postdose on Day 1 and on Days 2 (only in Cycle 1), 4, 5 (only in Cycle 1), 8, 12, 15, 19
Plasma Decay Half-Life (t1/2) of RO7051790 | Predose (0 hrs) on Day 1 of every cycle until end of treatment (up to 18 weeks, each cycle is 21 days); Cycles 1 and 2: 1, 2, 4, 6, 8 (only in Cycle 1) hrs postdose on Day 1 and on Days 2 (only in Cycle 1), 4, 5 (only in Cycle 1), 8, 12, 15, 19
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of RO7051790 | Predose (0 hrs) on Day 1 of every cycle until end of treatment (up to 18 weeks, each cycle is 21 days); Cycles 1 and 2: 1, 2, 4, 6, 8 (only in Cycle 1) hrs postdose on Day 1 and on Days 2 (only in Cycle 1), 4, 5 (only in Cycle 1), 8, 12, 15, 19
Area Under the Curve from Time Zero to End of Dosing Interval (AUCtau) of RO7051790 | Predose (0 hrs) on Day 1 of every cycle until end of treatment (up to 18 weeks, each cycle is 21 days); Cycles 1 and 2: 1, 2, 4, 6, 8 (only in Cycle 1) hrs postdose on Day 1 and on Days 2 (only in Cycle 1), 4, 5 (only in Cycle 1), 8, 12, 15, 19
Apparent Oral Clearance (CL/F) of RO7051790 | Predose (0 hrs) on Day 1 of every cycle until end of treatment (up to 18 weeks, each cycle is 21 days); Cycles 1 and 2: 1, 2, 4, 6, 8 (only in Cycle 1) hrs postdose on Day 1 and on Days 2 (only in Cycle 1), 4, 5 (only in Cycle 1), 8, 12, 15, 19
Apparent Volume of Distribution (Vz/F) of RO7051790 | Predose (0 hrs) on Day 1 of every cycle until end of treatment (up to 18 weeks, each cycle is 21 days); Cycles 1 and 2: 1, 2, 4, 6, 8 (only in Cycle 1) hrs postdose on Day 1 and on Days 2 (only in Cycle 1), 4, 5 (only in Cycle 1), 8, 12, 15, 19
Accumulation Ratio (RA) of RO7051790 | Predose (0 hrs) on Day 1 of every cycle until end of treatment (up to 18 weeks, each cycle is 21 days); Cycles 1 and 2: 1, 2, 4, 6, 8 (only in Cycle 1) hrs postdose on Day 1 and on Days 2 (only in Cycle 1), 4, 5 (only in Cycle 1), 8, 12, 15, 19

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- University of Alabama at Birmingham, Birmingham, Alabama, United States
- Canada (2):
  - The Ottawa Hospital Cancer Centre; Oncology, Ottawa, Ontario
  - University Health Network; Princess Margaret Hospital; Medical Oncology Dept, Toronto, Ontario
- Rigshospitalet; Onkologisk Klinik, København Ø, Denmark
- Institut Gustave Roussy, Villejuif, France
- Spain (3):
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Centro Integral Oncologico Clara Campal (CIOCC); Dirección Médica, Madrid